CLINICAL TRIAL: NCT06757777
Title: Evaluation of Remnant Cholesterol Levels and Monocyte-to-HDL-cholesterol Ratio As Predictors of Coronary Artery Disease Severity in Patients with Acute Coronary Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Isaac Ghaly Tawfik Girgis, Resident doctor, Assiut University
Other Study IDs: Monocyte to HDL Cholest. Ratio
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Acute Coronary Syndrome; ACS (acute Coronary Syndrome); Monocyte to HDL Cholesterol Ratio; STEMI; Non STEMI
Keywords: Acs; Acute coronary syndrome; STEMI; NON STEMI; Monocyte/HDL Ratio
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
1. Evaluation of serum level of remnant cholesterol and monocyte/HDL ratio as predictors of severity of coronary artery disease in patients with acute coronary syndrome.
2. Evaluate predictive value of remnant cholesterol serum level and monocyte/HDL ratio to detect in-hospital worse clinical outcomes and 45 days major adverse cardiac events (MACE) after acute coronary syndrome.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) refers to a group of conditions that include ST-elevation myocardial infarction (STEMI), non-ST elevation myocardial infarction (NSTEMI), and unstable angina. It is a type of coronary heart disease (CHD), ACS is the most common cause of death in patients with CAD and it is estimated that about 661,000 people in the United States suffer from ACS in 2016 ,which highlights the importance of risk assessment for ACS.

Elevated remnant cholesterol, including cholesterol carried in VLDL and chylomicron remnants, is emerging as a causal risk factor for ASCV in addition to elevated LDL-cholesterol ,Studies of the general population have shown that risk of myocardial infarction, ischemic stroke and peripheral artery disease is increased in individuals with elevated remnant cholesterol. High-density lipoprotein-cholesterol (HDL-C) exhibits anti-atherosclerotic effects by neutralizing the pro-inflammatory and pro-oxidant effects of monocytes via inhibiting the migration of macrophages and LDL oxidation in addition to the efflux of cholesterol from these cells. Furthermore, HDL plays a role in suppressing the activation of monocytes and proliferation-differentiation of monocyte progenitor cells. Thus, accumulation of monocytes and reduction of HDL-C may participate in atherosclerosis and cardiovascular diseases (CVD) .

Global Registry of Acute Coronary Events (GRACE) score is a risk assessment system for ACS based on risk factors summarized from clinical cases.

The Synergy between Percutaneous Coronary Intervention with Taxus and Cardiac Surgery (SYNTAX) score is a scoring system for risk stratification based on the anatomical characteristics of coronary artery lesions to help cardiologists, interventionists and surgeons to grade the complexity of coronary artery lesions .

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute coronary syndrome presented to ER of Assiut university hospital scheduled for primary PCI and able to provide informed consent.

Exclusion Criteria:

* Patients on previous statin therapy.
* Patients with severe renal dysfunction (creatinine clearance <30 mL/min) or other contraindications to PCI.
* Patients with missed data or who couldn't be followed up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome presented to ER of Assiut university hospital scheduled for primary PCI and able to provide informed consent
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-02-08 (Estimated); Primary Completion 2026-02-08 (Estimated); Study Completion 2026-03-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of serum level of remnant cholesterol and monocyte/HDL ratio as predictors of severity of coronary artery disease in patients with acute coronary syndrome. | Baseline

SECONDARY OUTCOMES:
Evaluate predictive value of remnant cholesterol serum level and monocyte/HDL ratio to detect in-hospital worse clinical outcomes and 45 days major adverse cardiac events (MACE) after acute coronary syndrome. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Isaac A Ghaly, Resident, Principal Investigator — Assiut University; Hanan A Mahmoud, Lecturer, Study Director — Assiut University; Khaled A Mohamed, Lecturer, Study Director — Assiut University

REFERENCES:
- [Background] Wadstrom BN, Wulff AB, Pedersen KM, Jensen GB, Nordestgaard BG. Elevated remnant cholesterol increases the risk of peripheral artery disease, myocardial infarction, and ischaemic stroke: a cohort-based study. Eur Heart J. 2022 Sep 7;43(34):3258-3269. doi: 10.1093/eurheartj/ehab705. PMID 34661640
- [Background] Zegre-Hemsey JK, Asafu-Adjei J, Fernandez A, Brice J. Characteristics of Prehospital Electrocardiogram Use in North Carolina Using a Novel Linkage of Emergency Medical Services and Emergency Department Data. Prehosp Emerg Care. 2019 Nov-Dec;23(6):772-779. doi: 10.1080/10903127.2019.1597230. Epub 2019 Apr 17. PMID 30885071